CLINICAL TRIAL: NCT02413762
Title: The Role of Gut Hormones and Hepcidin in Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Imperial College London Diabetes Centre (Other)
Responsible Party: Sponsor
Other Study IDs: IREC019
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- NGT, no insulin resistance: Individuals with normal glucose tolerance without a diagnosis of IGF, IGT or Diabetes Mellitus. No intervention.
- IFG/IGT/T2DM: Individuals with a diagnosis of impaired glucose tolerance, impaired fasting glucose or type 2 diabetes mellitus. No intervention.
- Insulin resistance without IGT: e.g. polycystic ovarian syndrome. No intervention.
- IGT, no insulin resistance: e.g. T1DM. No intervention.
- Previous metabolic surgery: Previous metabolic surgery for weight loss or treatment of T2DM. No intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention
  Groups: Previous metabolic surgery

SUMMARY:
This study aims to investigate the potential of the gut hormones GLP-1, PP, PYY and the iron regulatory hormone hepcidin as biomarkers for progression to complications in diabetes mellitus.

DETAILED DESCRIPTION:
Iron overload and mechanisms inducing insulin resistance are reciprocally linked. Dietary iron absorption, and iron uptake in liver and adipose tissue, are regulated through the hormone hepcidin. Iron is implicated in microvascular and macrovascular disease pathways and therefore hepcidin may represent a biomarker for progression to complications in type 2 diabetes mellitus.

Serum pancreatic polypeptide levels correlate with visceral adiposity and may therefore contribute to the diagnosis of, and risk stratification in, the metabolic syndrome.

Hypothesis:

Measuring iron status, incretin hormones and serum pancreatic polypeptide will facilitate discrimination of patients at risk of vascular complications of T2DM and clinically significant non-alcoholic fatty liver disease.

Statistical analysis:

Serum/plasma level of hormone under investigation corrected for age, sex, BMI, diabetes duration, blood pressure, lipid profile, smoking status, treatment for diabetes, hypertension and dyslipidaemia, and HbA1c using multinomial logistic regression and Cox regression models.

ELIGIBILITY:
Inclusion Criteria:

* all

Exclusion Criteria:

* lack of capacity for informed consent; vulnerable individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults resident in the UAE, attending ICLDC for normal healthcare.
Sampling Method: Non-Probability Sample
Enrollment: 1512 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Microvascular complication of diabetes mellitus - prevalence and incidence | 5 years
  Prevalence at enrolment and subsequent incidence of background diabetic retinopathy, preproliferative or proliferative retinopathy, or diabetic maculopathy; microalbuminuria defined as two episodes > 3 months apart of ACR > 2.5 (male) or > 3.5 (female) mg/umol. Assessed through patient recall and examination of electronic medical record.
Macrovascular complication of diabetes mellitus - prevalence and incidence | 5 years
  Prevalence at enrolment and subsequent incidence of composite endpoint of coronary artery disease (MI, ACS, percutaneous intervention), cerebrovascular disease (CVA, TIA), and peripheral arterial disease (ischaemic peripheral ulcer, revascularisation procedure, amputation). Assessed through patient recall and examination of electronic medical record.

SECONDARY OUTCOMES:
Progression to NAFLD or NASH | 5 years
  As defined by ultrasound criteria of NAFLD or evidence of fibrosis as measured using transient elastography, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Nader Lessan, MBBS FRCP MD, Principal Investigator — Imperial College London Diabetes Centre
Locations (1):
- Imperial College London Diabetes Centre, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Background] Sam AH, Sleeth ML, Thomas EL, Ismail NA, Mat Daud N, Chambers E, Shojaee-Moradie F, Umpleby M, Goldstone AP, Le Roux CW, Bech P, Busbridge M, Laurie R, Cuthbertson DJ, Buckley A, Ghatei MA, Bloom SR, Frost GS, Bell JD, Murphy KG. Circulating pancreatic polypeptide concentrations predict visceral and liver fat content. J Clin Endocrinol Metab. 2015 Mar;100(3):1048-52. doi: 10.1210/jc.2014-3450. Epub 2014 Dec 9. PMID 25490276
- [Background] Sam AH, Busbridge M, Amin A, Webber L, White D, Franks S, Martin NM, Sleeth M, Ismail NA, Daud NM, Papamargaritis D, Le Roux CW, Chapman RS, Frost G, Bloom SR, Murphy KG. Hepcidin levels in diabetes mellitus and polycystic ovary syndrome. Diabet Med. 2013 Dec;30(12):1495-9. doi: 10.1111/dme.12262. Epub 2013 Aug 19. PMID 23796160
- [Background] Fleming RE. Iron and inflammation: cross-talk between pathways regulating hepcidin. J Mol Med (Berl). 2008 May;86(5):491-4. doi: 10.1007/s00109-008-0349-8. No abstract available. PMID 18425494
- [Background] Fargion S, Dongiovanni P, Guzzo A, Colombo S, Valenti L, Fracanzani AL. Iron and insulin resistance. Aliment Pharmacol Ther. 2005 Nov;22 Suppl 2:61-3. doi: 10.1111/j.1365-2036.2005.02599.x. PMID 16225476
- [Background] Semple RK, Sleigh A, Murgatroyd PR, Adams CA, Bluck L, Jackson S, Vottero A, Kanabar D, Charlton-Menys V, Durrington P, Soos MA, Carpenter TA, Lomas DJ, Cochran EK, Gorden P, O'Rahilly S, Savage DB. Postreceptor insulin resistance contributes to human dyslipidemia and hepatic steatosis. J Clin Invest. 2009 Feb;119(2):315-22. doi: 10.1172/JCI37432. Epub 2009 Jan 26. PMID 19164855